CLINICAL TRIAL: NCT00566241
Title: An Investigation Into the Use of IGF-1 Therapy in Patients With Cystic Fibrosis
Brief Title: IGF-1 Therapy in Patients With Cystic Fibrosis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Insufficient recruitment
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Thomas A. Wilson, Professor of Pediatrics, Stony Brook University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IGF-1 in Cystic Fibrosis
Record Dates: First submitted 2007-11-30; First posted 2007-12-03 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Cystic Fibrosis
Keywords: Body weight; Body composition; Pulmonary function; Carbohydrate tolerance
MeSH Terms: conditions — Cystic Fibrosis; Body Weight | interventions — mecasermin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IGF-1 (Experimental): Recombinant human IGF-1
  Interventions: Drug: recombinant human IGF-1
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: recombinant human IGF-1 — rhIGF-1
  Other Names: mecasermin
  Arms: IGF-1
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
28 week pilot study to examine the efficacy of recombinant human IGF-1 on body weight and composition in adults with cystic fibrosis.

DETAILED DESCRIPTION:
28 week, double blind, cross over study to determine the efficacy of rhIGF-1 on body weight and body composition in patients with cystic fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cystic fibrosis as proven by either sweat chloride or DNA analysis.
* Age >= 18 yr.
* Tanner stage: Femake Breasts: 4-5 Male Genitalia: 4-5

Exclusion criteria:

* Hemoglobin A1C > 8.5 %
* Diabetic retinopathy
* Obstructive sleep apnea
* Respiratory failure requiring mechanical ventilation.
* Status post pulmonary transplantation.
* Concurrent or recent (within past 6 months) receipt of human growth hormone.
* History of adverse side effects to growth hormone other than carbohydrate intolerance.
* Pregnancy or attempting pregnancy.
* Women who are breast feeding.
* Sexually active women who refuse to use or are incapable of responsibly using reliable contraception.
* Proven non compliance with medical regimens.
* Inability or refusal to take subcutaneous injections.
* Known allergy to components in the IGF-I preparation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2008-06; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Body weight and body composition | 28 weeks

SECONDARY OUTCOMES:
Pulmonary function | 28 weeks
Carbohydrate tolerance | 28 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Thomas A Wilson, MD, Principal Investigator — State Univeristy of New York, Stony Brook, NY
Locations (1):
- State University of New York, Stony Brook, New York, United States